CLINICAL TRIAL: NCT02037815
Title: Correlation of Measured and Calculated Serum Osmolality During Mannitol or Hypertonic Saline Infusion in Patients After Craniotomy
Brief Title: Correlation of Measured and Calculated Serum Osmolality During Hyperosmolar Drugs Infusion in Patients After Craniotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: KY-2013-002-003
Record Dates: First submitted 2014-01-13; First posted 2014-01-16 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Brain Edema
Keywords: hyperosmolar drugs; mannitol; hypertonic saline; serum osmolality; correlation
MeSH Terms: conditions — Brain Edema | interventions — Infusions, Intravenous; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Mannitol (Experimental): 20% mannitol solution, 125 ml, IV infusion in 15 min
  Interventions: Drug: 20% mannitol solution, 125 ml, IV infusion in 15 min
- Hypertonic saline (Experimental): 3.1% sodium chloride solution, 125 ml, IV infusion in 15 min
  Interventions: Drug: 3.1% sodium chloride solution, 125 ml, IV infusion in 15 min

INTERVENTIONS:
Drug: 20% mannitol solution, 125 ml, IV infusion in 15 min
  Arms: Mannitol
Drug: 3.1% sodium chloride solution, 125 ml, IV infusion in 15 min
  Arms: Hypertonic saline

SUMMARY:
Osmotherapy has been used as the medical treatment for brain edema and intracranial hypertension in critically brain injured patients. Measurement of serum osmolality during osmotherapy is of clinical importance to determine clinical efficacy, adjust dosage and avoid side effect. Serum osmolality is often measured in laboratory by cryoscopic technique as the reference method. However, in clinical setting, routine measurement of serum osmolality is not feasible at bedside, either in intensive care unit (ICU) or neurosurgical ward. Therefore, clinicians usually estimate serum osmolality by using equations derived from serum osmoles that can be measured by bedside blood gas analysis or routine laboratory chemical analysis, such as sodium, potassium, urea, and glucose. In present study, mannitol or hypertonic saline will be used in patients after craniotomy, and serum osmolality will be measured before and during drug infusion. Investigators hypothesize that the correlation of measured and calculated serum osmolality is better during infusion of hypertonic saline than mannitol.

ELIGIBILITY:
Inclusion Criteria:

* adult patients after elective craniotomy, requiring hyperosmolar agents for prevention or treatment of brain edema

Exclusion Criteria:

* age younger than 18 yr or older than 65 yr
* history of diabetes
* unstable hemodynamic condition
* presence of renal failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Difference between the measured and calculated serum osmolality. | Immediately before the infusion of mannitol and hypertonic saline, and 15, 30, 60, 120, 240, and 360 minutes after the administration of the study drugs

SECONDARY OUTCOMES:
Serum osmolality | Immediately before the infusion of mannitol and hypertonic saline, and 15, 30, 60, 120, 240, and 360 minutes after the administration of the study drugs
Concentration of serum sodium | Immediately before the infusion of mannitol and hypertonic saline, and 15, 30, 60, 120, 240, and 360 minutes after the administration of the study drugs

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Principal Investigator — Neurosurgical ICU, Beijing Tiantan Hospital, Capital Medical University
Locations (1):
- Neurosurgical ICU, Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li Q, Chen H, Hao JJ, Yin NN, Xu M, Zhou JX. Agreement of measured and calculated serum osmolality during the infusion of mannitol or hypertonic saline in patients after craniotomy: a prospective, double-blinded, randomised controlled trial. BMC Anesthesiol. 2015 Oct 7;15:138. doi: 10.1186/s12871-015-0119-4. PMID 26445777
- [Derived] Li Q, Xu M, Zhou JX. Correlation of measured and calculated serum osmolality during mannitol or hypertonic saline infusion in patients after craniotomy: a study protocol and statistical analysis plan for a randomised controlled trial. BMJ Open. 2014 Apr 23;4(4):e004921. doi: 10.1136/bmjopen-2014-004921. PMID 24760352